CLINICAL TRIAL: NCT03807934
Title: Cerebral Excitability and Cognitive Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Tad Brunye, PI, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1303018
Record Dates: First submitted 2019-01-11; First posted 2019-01-17 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Cognitive Change
Keywords: transcranial direct current stimulation; cognitive psychology; noninvasive brain stimulation; electrical brain stimulation

STUDY DESIGN:
Intervention Model Description: Repeated-measures crossover design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active High-Definition Stimulation (Experimental): Active high-definition stimulation of targeted brain regions involved in perception and cognition.
  Interventions: Other: Stimulation via Soterix Medical or Neuroelectrics noninvasive brain stimulation systems
- Sham High-Definition Stimulation (Sham Comparator): Sham high-definition stimulation of targeted brain regions involved in perception and cognition.
  Interventions: Other: Stimulation via Soterix Medical or Neuroelectrics noninvasive brain stimulation systems

INTERVENTIONS:
Other: Stimulation via Soterix Medical or Neuroelectrics noninvasive brain stimulation systems — Active (at or below 2mA) versus sham (at or below 0.5mA) stimulation targeting brain regions engaged during verbal and/or spatial perceptual and cognitive processing. Brain stimulation devices are not currently regulated by the United States Food and Drug Administration. Local IRB has determined the devices to be non-significant risk (NSR) devices via abbreviated investigational device exemption (IDE) procedure.

SUMMARY:
This study investigates the perceptual and cognitive influences of low-intensity electrical brain stimulation (transcranial direct current stimulation; tDCS), versus control (sham) conditions.

ELIGIBILITY:
Inclusion Criteria:

- Between ages of 18-65.

Exclusion Criteria:

* History of adverse reaction to tDCS (trans-cranial direct current stimulation).
* History of seizure activity.
* History of head injury (including neurosurgery).
* History of illness causing brain injury.
* History of other brain-related condition (such as traumatic brain injury).
* History of diagnosis with a neurological or psychiatric disorder.
* History of metal in head (outside of mouth), such as shrapnel, surgical clips, or fragments from welding or metalwork.
* History of sensitive scalp.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2013-04-15 (Actual); Primary Completion 2023-04-14 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
Visual perceptual performance | 36 weeks
  Ability to accurately and efficiently perceive perceptual information, including threat detection, local contrast gradient detection, face memory, and intent appraisal. All are computerized tasks.
Verbal cognitive performance | 36 weeks
  Ability to accurately and efficiently process verbal information, including verbal cued free association tasks, verbal long-term memory, and language comprehension. All are computerized tasks.
Spatial cognitive performance | 72 weeks
  Ability to accurately and efficiently process spatial information, including map learning, virtual urban navigation, and mental rotation. All are computerized tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Result] Brunye TT, Hussey EK, Fontes EB, Ward N. Modulating Applied Task Performance via Transcranial Electrical Stimulation. Front Hum Neurosci. 2019 Apr 30;13:140. doi: 10.3389/fnhum.2019.00140. eCollection 2019. PMID 31114491
- [Result] Brunye TT, Smith AM, Horner CB, Thomas AK. Verbal long-term memory is enhanced by retrieval practice but impaired by prefrontal direct current stimulation. Brain Cogn. 2018 Dec;128:80-88. doi: 10.1016/j.bandc.2018.09.008. Epub 2018 Nov 8. PMID 30414699
- [Result] Brunye TT. Modulating Spatial Processes and Navigation via Transcranial Electrical Stimulation: A Mini Review. Front Hum Neurosci. 2018 Jan 9;11:649. doi: 10.3389/fnhum.2017.00649. eCollection 2017. PMID 29375346
- [Result] Brunye TT, Moran JM, Cantelon J, Holmes A, Eddy MD, Mahoney CR, Taylor HA. Increasing breadth of semantic associations with left frontopolar direct current brain stimulation: a role for individual differences. Neuroreport. 2015 Mar 25;26(5):296-301. doi: 10.1097/WNR.0000000000000348. PMID 25714417
- [Result] Brunye TT, Holmes A, Cantelon J, Eddy MD, Gardony AL, Mahoney CR, Taylor HA. Direct current brain stimulation enhances navigation efficiency in individuals with low spatial sense of direction. Neuroreport. 2014 Oct 22;25(15):1175-9. doi: 10.1097/WNR.0000000000000214. PMID 25144391